CLINICAL TRIAL: NCT04441502
Title: Identification of Predictors for the Evolution of COVID-19 Related Interstitial Pneumonia by Transcriptomic and Seroproteomic Techniques
Brief Title: Identification of Predictors for the Evolution of COVID-19 Related Pneumonia by Transcriptomic and Seroproteomic
Acronym: COVID_OMICS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Marco Ranucci, Head of Cardiothoracic and Vascular Anesthesia and Intensive Care, IRCCS Policlinico S. Donato
Other Study IDs: COVID19_OMICS
Record Dates: First submitted 2020-06-12; First posted 2020-06-22 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Covid19; Interstitial Pneumonia
Keywords: inflammation; thrombin generation; fibrinogenesis; fibrinolysis
MeSH Terms: conditions — COVID-19; Lung Diseases, Interstitial; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, whole blood, PBMC samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigating group aims at performing an observational, prospective study that involves the evaluation of circulating biomarkers predictive of clinical evolution in patients suffering from COVID-19 disease.

In particular, the aim will be to verify whether there are transcripts or cytokines / chemokines in peripheral blood, modulated differently in patients with COVID-19, distinguished on the basis of the evolution towards more severe clinical pictures that require patient intubation or that show signs of cardiovascular damage.

The study will be based on the transcriptional analysis of the entire genome and serum protein to evaluate the expression of a broad spectrum of cytokines and chemokines. Genome analysis will allow the genotype to be correlated to the identified gene expression profiles.

DETAILED DESCRIPTION:
Study design This observational, prospective, monocentric study will make use of the recruitment of consecutive patients with COVID-19. Enrollment will last 6 months or, considering the desirable drop in infections in the next few weeks, until exhaustion of enrolled patients. Enrollment will be followed by 18 months dedicated to transcriptomics and seroproteomics investigations, for a total duration of the study of 24 months.

All patients will receive optimal medical therapy, and will undergo laboratory or instrumental examinations (chest x-ray, CT, echocardiography) as needed.

Blood samples will be taken at the entrance and then twice a week for the duration of the hospitalization (generally 2-3 weeks).

Anamnesis will be noted for all patients. In addition, at all times, patients will undergo clinical evaluation and the following laboratory tests, which include:

* blood count
* biochemistry
* standard coagulation and thrombin generation, fibrin generation and fibrinolysis (INR, PTT, D-dimer, Tissue Plasminogen Activator TPA, Plasminogen Activator Inhibitor PAI-2, Plasmin-AntiPlasmin complex PAP, Thrombin activated Fibrinolysis Inhibitor TAFI, Thrombin-AntiThrombin complex TAT, Prothrombin Fragment PF 1+2, Fibrinopeptide A)
* inflammation/infection (IL-6, procalcitonin, ferritin, PCR, sCD14, TLR3 and 4, RANTES, CCR3 and 4
* other (troponin I, NT-pro-BNP, Hb1Ac). A subgroup of patients will undergo a microcirculation analysis with SDF (Sidestream Dark Field imaging).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Positivity to the test for SARS-Cov-2
3. Informed consent to enrollment in the study.
4. For Intensive Care patients: entry into the intensive unit and / or endotracheal intubation for no more than 4 days.
5. For patients in the COVID19 wards: home hospitalization or emergency room for no more than 4 days.

Exclusion Criteria:

1. Age less than 18 years
2. Pregnant women
3. Patients with malignant neoplasm, autoimmune diseases.
4. Hospitalization as transfer from another hospital or other similar facility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 240 patients with COVID-19 will be recruited, including up to 60 patients from the intensive care and 180 from the specialized COVID19 departments of the IRCCS Policlinico San Donato. The sample size is estimated based on the average length of hospitalization of the patients and the maximum capacity of the clinical and laboratory units involved in the study.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Circulating markers for COVID-19 signature | From ICU/ward admission for 8 weeks follow/up
  Identify circulating transcripts (coding and non-coding for proteins) or cytokines and chemokines which, alone or in combination (COVID19_signature), are predictive of adverse events (death, endotracheal intubation) and the prognostic capacity of COVID19_signature in the prediction of adverse events in additional to the use of standard clinical parameters

SECONDARY OUTCOMES:
COVID-19 signature and adverse cardiovascular events | From ICU/ward admission for 8 weeks follow/up
  Evaluate the association of COVID19_signature with adverse cardiovascular events. Adverse cardiovascular events are defined: death from cardiovascular causes, acute coronary syndrome, troponin T levels greater than the ninety-ninth percentile of the upper reference limit, stroke, cardiac arrhythmias, development of heart failure, venous thromboembolism
COVID-19 related coagulation pattern | From ICU/ward admission for 8 weeks follow/up
  Evaluate, in a subset of 20 patients, the characteristics of the coagulation pattern with specific tests for thrombin generation and fibrinolysis.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ranucci, MD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yin Y, Wunderink RG. MERS, SARS and other coronaviruses as causes of pneumonia. Respirology. 2018 Feb;23(2):130-137. doi: 10.1111/resp.13196. Epub 2017 Oct 20. PMID 29052924
- [Background] Xu J, Zhao S, Teng T, Abdalla AE, Zhu W, Xie L, Wang Y, Guo X. Systematic Comparison of Two Animal-to-Human Transmitted Human Coronaviruses: SARS-CoV-2 and SARS-CoV. Viruses. 2020 Feb 22;12(2):244. doi: 10.3390/v12020244. PMID 32098422
- [Background] Chen Y, Liu Q, Guo D. Emerging coronaviruses: Genome structure, replication, and pathogenesis. J Med Virol. 2020 Apr;92(4):418-423. doi: 10.1002/jmv.25681. Epub 2020 Feb 7. PMID 31967327
- [Background] Ren LL, Wang YM, Wu ZQ, Xiang ZC, Guo L, Xu T, Jiang YZ, Xiong Y, Li YJ, Li XW, Li H, Fan GH, Gu XY, Xiao Y, Gao H, Xu JY, Yang F, Wang XM, Wu C, Chen L, Liu YW, Liu B, Yang J, Wang XR, Dong J, Li L, Huang CL, Zhao JP, Hu Y, Cheng ZS, Liu LL, Qian ZH, Qin C, Jin Q, Cao B, Wang JW. Identification of a novel coronavirus causing severe pneumonia in human: a descriptive study. Chin Med J (Engl). 2020 May 5;133(9):1015-1024. doi: 10.1097/CM9.0000000000000722. PMID 32004165
- [Background] Yan R, Zhang Y, Li Y, Xia L, Guo Y, Zhou Q. Structural basis for the recognition of SARS-CoV-2 by full-length human ACE2. Science. 2020 Mar 27;367(6485):1444-1448. doi: 10.1126/science.abb2762. Epub 2020 Mar 4. PMID 32132184
- [Background] Liu J, Zheng X, Tong Q, Li W, Wang B, Sutter K, Trilling M, Lu M, Dittmer U, Yang D. Overlapping and discrete aspects of the pathology and pathogenesis of the emerging human pathogenic coronaviruses SARS-CoV, MERS-CoV, and 2019-nCoV. J Med Virol. 2020 May;92(5):491-494. doi: 10.1002/jmv.25709. Epub 2020 Feb 21. PMID 32056249
- [Background] Ranucci M, Ballotta A, Di Dedda U, Baryshnikova E, Dei Poli M, Resta M, Falco M, Albano G, Menicanti L. The procoagulant pattern of patients with COVID-19 acute respiratory distress syndrome. J Thromb Haemost. 2020 Jul;18(7):1747-1751. doi: 10.1111/jth.14854. Epub 2020 May 6. PMID 32302448
- [Background] Fung SY, Yuen KS, Ye ZW, Chan CP, Jin DY. A tug-of-war between severe acute respiratory syndrome coronavirus 2 and host antiviral defence: lessons from other pathogenic viruses. Emerg Microbes Infect. 2020 Mar 14;9(1):558-570. doi: 10.1080/22221751.2020.1736644. eCollection 2020. PMID 32172672
- [Background] Keidar S, Kaplan M, Gamliel-Lazarovich A. ACE2 of the heart: From angiotensin I to angiotensin (1-7). Cardiovasc Res. 2007 Feb 1;73(3):463-9. doi: 10.1016/j.cardiores.2006.09.006. Epub 2006 Sep 19. PMID 17049503
- [Background] Zheng YY, Ma YT, Zhang JY, Xie X. COVID-19 and the cardiovascular system. Nat Rev Cardiol. 2020 May;17(5):259-260. doi: 10.1038/s41569-020-0360-5. PMID 32139904
- [Background] Kwong JC, Schwartz KL, Campitelli MA, Chung H, Crowcroft NS, Karnauchow T, Katz K, Ko DT, McGeer AJ, McNally D, Richardson DC, Rosella LC, Simor A, Smieja M, Zahariadis G, Gubbay JB. Acute Myocardial Infarction after Laboratory-Confirmed Influenza Infection. N Engl J Med. 2018 Jan 25;378(4):345-353. doi: 10.1056/NEJMoa1702090. PMID 29365305
- [Background] Nguyen JL, Yang W, Ito K, Matte TD, Shaman J, Kinney PL. Seasonal Influenza Infections and Cardiovascular Disease Mortality. JAMA Cardiol. 2016 Jun 1;1(3):274-81. doi: 10.1001/jamacardio.2016.0433. PMID 27438105
- [Background] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Peiris JS, Chu CM, Cheng VC, Chan KS, Hung IF, Poon LL, Law KI, Tang BS, Hon TY, Chan CS, Chan KH, Ng JS, Zheng BJ, Ng WL, Lai RW, Guan Y, Yuen KY; HKU/UCH SARS Study Group. Clinical progression and viral load in a community outbreak of coronavirus-associated SARS pneumonia: a prospective study. Lancet. 2003 May 24;361(9371):1767-72. doi: 10.1016/s0140-6736(03)13412-5. PMID 12781535
- [Background] Greco S, Gorospe M, Martelli F. Noncoding RNA in age-related cardiovascular diseases. J Mol Cell Cardiol. 2015 Jun;83:142-55. doi: 10.1016/j.yjmcc.2015.01.011. Epub 2015 Jan 29. PMID 25640162
- [Background] Carrara M, Fuschi P, Ivan C, Martelli F. Circular RNAs: Methodological challenges and perspectives in cardiovascular diseases. J Cell Mol Med. 2018 Nov;22(11):5176-5187. doi: 10.1111/jcmm.13789. Epub 2018 Sep 11. PMID 30277664
- [Background] Beermann J, Piccoli MT, Viereck J, Thum T. Non-coding RNAs in Development and Disease: Background, Mechanisms, and Therapeutic Approaches. Physiol Rev. 2016 Oct;96(4):1297-325. doi: 10.1152/physrev.00041.2015. PMID 27535639
- [Background] Zhao S, Li CI, Guo Y, Sheng Q, Shyr Y. RnaSeqSampleSize: real data based sample size estimation for RNA sequencing. BMC Bioinformatics. 2018 May 30;19(1):191. doi: 10.1186/s12859-018-2191-5. PMID 29843589
- See also: World Health Organization. Novel coronavirus (2019-nCoV) SITUATION REPORT - 1 21 JANUARY 2020 — https://www.who.int/docs/default-source/coronaviruse/situation-reports/20200121-sitrep-1-2019-ncov.pdf?sfvrsn=20a99c10_4